CLINICAL TRIAL: NCT07090213
Title: Turkish Version of Pelvi-Perineal Surgery Sexuality Questionnaire: Translation, Cultural Adaptation and Validation
Brief Title: Turkish Version of Pelvi-Perineal Surgery Sexuality Questionnaire
Status: Completed | Type: Observational
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Betül Çınar, Lecturer, PhD, Bezmialem Vakif University
Other Study IDs: bvubcinar03
Record Dates: First submitted 2025-07-21; First posted 2025-07-29 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Surgery; Maternal, Uterus or Pelvic Organs, Affecting Fetus
Keywords: validation; cultural adaptation; pelvic surgery

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Survey using a questionnaire — Eighty women, determined by the number of questions times the rule of 10, will be asked to fill out the Pelvi-Perineal Surgery Sexuality Questionnaire - PPSSQ and Female Sexual Function Index (FSFI) questionnaires and will be asked to fill out the PPSSQ again 7 days later for test-retest reliability.
  Other Names: Permission was obtained from the original owner of Pelvi-Perineal Surgery Sexuality Questionnaire - PPSSQ for the Turkish cultural adaptation, validity and reliability study.

SUMMARY:
This prospective, multicentre observational study translates the 13-item Pelvi-Perineal Surgery Sexuality Questionnaire (PPSSQ) from French to Turkish, culturally adapts it, and evaluates its reliability, validity and responsiveness in Turkish-speaking women covering from pelvic floor surgery.

DETAILED DESCRIPTION:
Sexual function is a key outcome after incontinence or prolapse surgery; however, no Turkish tool specifically captures surgery-related sexual issues. The Pelvi-Perineal Surgery Sexuality Questionnaire (PPSSQ) was recently validated in France and measures two dimensions ("Sexual Health" and "Discomfort & Pain") with good psychometric performance.

The English version of PPSSQ will be adapted for Turkish use according to the established guidelines for cross-cultural adaptation of self-reported questionnaires. The guideline has 5 steps: (1) translation, (2) synthesis, (3) back translation, (4) evaluation by a team of experts, and (5) pretests. 80 sexually active and inactive women (≥18 y) with mid-urethral sling, vaginal or laparoscopic prolapse repair (with/without mesh) will be recruited. Participants will complete the Turkish version of the Female Sexual Function Index (FSFI-Turkish) on the first visit and again 7 days later for validation purposes. Internal consistency will be tested using Cronbach's alpha, and the test-retest reliability will be assessed by calculating the intra-class correlation coefficient.

ELIGIBILITY:
Inclusion Criteria:

* Having had pelvic surgery more than 12 months ago
* Being sexually active for the last three months
* Being literate

Exclusion Criteria:

* Not having had a sexual partner for at least three months
* Receiving anti-estrogen therapy for any reason
* Having a history of gynecological or breast cancer
* Not understanding written Turkish

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — No. Participant eligibility is based on assigned sex at birth (biological female).
Study Population: Women who have had pelvic surgery more than 12 months ago and have been sexually active for the past three months.
Sampling Method: Non-Probability Sample
Enrollment: 113 (Actual)
Dates: Start 2025-07-22 (Actual); Primary Completion 2025-11-05 (Actual); Study Completion 2026-01-05 (Actual)

PRIMARY OUTCOMES:
Pelvi-Perineal Surgery Sexuality Questionnaire | 1 week
  The Pelvi-Perineal Surgery Sexuality Questionnaire (PPSSQ) is a 13-question self-questionnaire validated in a population of sexually active women or not, operated on for stress urinary incontinence or pelvic organ prolapse by laparoscopy or vaginal surgery, with or without mesh. The domains are "Sexual Health" and "Discomfort and Pain." The questionnaire is calculated out of 100 points, with a higher score indicating better sexual function.

SECONDARY OUTCOMES:
Female Sexual Function Index (FSFI) | 1 week
  It is a 19-item multidimensional self-reporting measure that quantified female sexual dysfunction in six domains: desire, arousal, lubrication, orgasm, satisfaction, and pain. These questions ask about patients' sexual feelings and responses during the past 4 weeks. FSFI use a 5-point Likert scale ranging from 1-5 with higher scores indicating greater levels of sexual functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Betul Cinar, PhD, Principal Investigator — Bezmialem Vakif University
Locations (1):
- Bezmialem Vakif University, Istanbul, Turkey (Türkiye)